CLINICAL TRIAL: NCT05281211
Title: Nutrition and EXercise Prehabilitation to Reduce Morbidity (NEXPREM) Following Major Liver Surgery in Sarcopenic Patients
Brief Title: Nutrition and Exercise Prehabilitation to Reduce Morbidity Following Major Liver Surgery in Sarcopenic Patients
Acronym: NEXPREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Camillo Hospital, Rome (Other)
Responsible Party: Principal Investigator, Giammauro Berardi, Principal Investigator, San Camillo Hospital, Rome
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022.01
Record Dates: First submitted 2022-02-12; First posted 2022-03-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Liver Cancer; Surgery; Sarcopenia
Keywords: sarcopenia; liver cancer; liver surgery; hepatectomy
MeSH Terms: conditions — Liver Neoplasms; Sarcopenia | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative Nutrition+Exercise (Experimental): Preoperative nutrition and exercise pre-habilitation followed by major liver resection.
  Interventions: Dietary Supplement: Nutrition; Behavioral: Exercise
- Upfront Surgery (No Intervention): Upfront major liver resection.

INTERVENTIONS:
Dietary Supplement: Nutrition — 6 weeks nutrition implementation in the form of branched chain amino acids and immune-system boosters twice daily for 4 weeks and once daily for 2 weeks
  Arms: Preoperative Nutrition+Exercise
Behavioral: Exercise — 6 weeks exercise 30 minutes' walk/day or 2000 extra steps daily
  Arms: Preoperative Nutrition+Exercise

SUMMARY:
NEXPREM is a single-center non-blinded randomized controlled trial investigating preoperative exercise and nutrition for sarcopenic patients in major hepatic surgery for liver malignancies. Patients with sarcopenia undergoing major hepatectomies have high rates of postoperative complications. Previous studies have demonstrated that preoperative rehabilitation with exercise and nutrition may help reduce the negative impact of sarcopenia. The investigator's hypothesis is that preoperative nutrition and exercise may reduce complications in sarcopenic patients undergoing major hepatectomies. Sarcopenic patients at diagnosis will be randomized in Group A undergoing upfront surgery and Group B undergoing preoperative rehabilitation. Outcome will be overall 90 day morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age >18.
* Sarcopenic patients diagnosed by both qualitative and quantitative analysis.
* Patients with primary or secondary liver malignancies.
* Patients undergoing major liver resections intended as 3 or more contiguous segments
* Patients undergoing open, laparoscopic, or robotic resections.

Exclusion Criteria:

* Minor liver resections intended as less than 3 contiguous segments.
* Patients with intrahepatic, hilar, or extrahepatic cholangiocarcinomas.
* Patients with liver tumors for whom 6 weeks interval from diagnosis to surgery could not be waited (i.e., large HCCs on healthy livers not requiring preoperative portal vein occlusion, CRLM without preoperative administration of anti-VEGF drug who therefore do not require 6 weeks of chemotherapy washout)
* Patients with benign liver lesions.
* Patients undergoing extrahepatic liver resections.
* Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy (ALPPS) procedure.
* Patients with physical disabilities, unable to exercise.
* Patients with inadequate kidney function.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing 90 day morbidity | 90 days
  Patients experiencing complications within 90 days of surgery

SECONDARY OUTCOMES:
Number of participants experiencing 90 days postoperative major complications according to Clavien-Dindo classification | 90 days
Number of participants experiencing 90 days postoperative mortality. | 90 days
Number of participants being readmitted within 90 days of surgery. | 90 days
Number of participants being Sarcopenic after 6 weeks of prehabilitation. | 6 weeks
Number of participants Alive ( Overall Survival) | 3 years
Number of participants being disease free (Disease free survival) | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - San Camillo Hospital, Rome, Italy
  - San Camillo Forlanini, Roma, RM

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Berardi G, Cucchetti A, Colasanti M, Angrisani M, Moschetta G, Chiappori D, Marini A, Antonelli G, Ferretti S, Meniconi RL, Guglielmo N, Mariano G, Usai S, Ettorre GM. Prehabilitation With Exercise and Nutrition to Reduce Morbidity of Major Hepatectomy in Patients With Sarcopenia: The PREHEP Randomized Clinical Trial. JAMA Surg. 2025 Oct 1;160(10):1068-1075. doi: 10.1001/jamasurg.2025.3102. PMID 40864449